CLINICAL TRIAL: NCT00059618
Title: A Phase I Study Evaluating the Safety and Tolerability of PS-341(Bortezomib)and Carboplatin in Patients With Platinum- and Taxane-Resistant Recurrent Ovarian Cancer, Primary Peritoneal Cancer, and Fallopian Tube Cancer
Brief Title: PS-341 Plus Carboplatin in Platinum and Taxane Resistant Recurrent Ovarian Cancer, Primary Peritoneal Cancer, and Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-114
Record Dates: First submitted 2003-04-29; First posted 2003-04-30 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Platinum Resistant; Taxane Resistant; Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer; Bortezomib; PS-341; Velcade; LDP-341; MLN341; Carboplatin; Paraplatin
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bortezomib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib (Experimental): PS-341 (Bortezomib) 0.8-1.5 mg/m^2 IV push + Carboplatin (AUC 5) IV on Day 1 of each cycle, then Bortezomib alone on Days 4, 8 and 11 in each 28 day cycle.
  Interventions: Drug: PS-341 (Bortezomib); Drug: Carboplatin

INTERVENTIONS:
Drug: PS-341 (Bortezomib) — Starting dose 0.8 mg/m^2 given by vein over 5-10 seconds Day 1, 4, 8 and 11 of 28 day cycle for 8 cycles.
  Other Names: Velcade; LDP-341; MLN341
Drug: Carboplatin — AUC 5 by vein administered over one hour Day 1 of 28 day cycle for 8 cycles.
  Other Names: Paraplatin

SUMMARY:
The goal of this clinical research study is to find the highest safe dose of PS-341 that can be given with carboplatin chemotherapy as a treatment for patients with ovarian, abdominal, or fallopian tube cancer. Researchers also hope to find out if giving these drugs together will help shrink or slow the growth of tumors in patients who are considered resistant to platinum drugs. The safety of these drugs will also be studied.

DETAILED DESCRIPTION:
Bortezomib is a drug that turns off certain genes and proteins inside the cancer cell that are responsible for cell growth. Researchers believe that when certain genes and proteins are turned off, the ability of the cancer cell to survive is decreased.

Before treatment starts, participants will have a complete checkup, blood tests, a urine test, a heart test, a chest x-ray, and either a CT scan or MRI scan. Women able to have children must have a negative blood pregnancy test within 14 days of beginning treatment. Blood tests and a complete checkup will also be done before each course of therapy and a month after treatment ends. Approximately 2-3 teaspoons of blood will be obtained for routine blood tests each time blood is drawn during this study.

Participants in this study will receive Bortezomib and carboplatin through a catheter (tube) placed in a vein. This is Day 1 of therapy. Bortezomib is given first (over 5 to 10 seconds) followed by carboplatin (over one hour). Bortezomib is then given alone on Days 4, 8, and 11. There is no treatment given on Days 12-28. One course of therapy is 28 days long and includes one dose of carboplatin and 4 doses of Bortezomib. All treatment is given on an outpatient basis at M. D. Anderson.

There are 4 different dose levels of Bortezomib being studied. The dose of Bortezomib that participants receive will depend on when they are enrolled. It will also depend on whether or not other participants had side effects from their treatment. Up to 6 patients could be treated at each dose.

Before each course of therapy, participants will have a physical exam and blood tests. A CT scan or MRI scan is repeated after Cycles 2 and 4 and at the end of treatment. Participants who have a partial or complete response (the tumor shrinks by more than 50% or disappears completely) will have a repeat CT or MRI 4 weeks later to confirm the response.

Participants may receive up to 8 courses of treatment. If the disease gets worse or if intolerable side effects occur, participants will be taken off study.

This is an investigational study. Bortezomib is approved for use by the FDA, in patients with multiple myeloma. Carboplatin is approved by the FDA, though its use with Bortezomib is experimental. A total of 24 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed ovarian cancer, primary peritoneal cancer, or fallopian tube cancer with advanced and/or metastatic disease. All patients must be considered platinum- and taxane- resistant.
* Platinum resistance is defined as:

  1. Progression of disease during platinum or taxane chemotherapy, or
  2. Progression of disease within 6 months of completing platinum or taxane chemotherapy
  3. Failure to achieve a complete response, with persistent macroscopic disease, after 6 cycles of chemotherapy, if the last two cycles had no measurable change in disease status
* Patients may have had any number of prior chemotherapy regimens, except high dose chemotherapy an/or peripheral blood stem cell transplantation (high dose: higher than the standard doses of chemotherapy)
* Patients must have measurable disease.
* Zubrod performance status of < 2.
* Patients must give voluntary written informed consent before performance of any study-related procedure not part of normal medical care.
* Adequate liver, renal and bone marrow function, defined as:

  * Absolute neutrophil count (ANC) > 1.5 x 10^9/L.
  * Platelets > 100 x 10^9/L
  * Total bilirubin < 1.7 umol/L
  * Alanine transaminase (ALT) and aspartate transaminase (AST) < 1.5 x Upper Limits of Normal (ULN)
  * Alkaline phosphatase < 2.5 x ULN.
  * Serum creatinine < 1.5 x ULN.

Exclusion Criteria:

* Chemotherapy within four weeks of first course of PS-341. (Patients may have been on hormonal therapy).
* Patients who previously received high-dose chemotherapy (higher than the standard doses of chemotherapy) and/or peripheral blood stem cell transplantation.
* Radiation therapy within four weeks of enrollment (excepting palliative XRT).
* Patients not recovered from toxic effects of previous chemotherapy, radiation therapy, or antibody therapy.
* Patients with > Grade 2 peripheral neuropathy.
* Surgery within four weeks of study enrollment.
* History of severe hypersensitivity reaction to carboplatin
* Electrocardiographic evidence of acute ischemia or new conduction system abnormalities.
* Myocardial infarction within six months of enrollment.
* Patients with brain metastases or central nervous system disease as evidenced by clinical symptoms.
* History of other malignancy, except nonmelanoma skin cancer or carcinoma in-situ of the cervix, unless in complete remission and off all therapy for that disease for a minimum of 5 years. Chemotherapy given for prior cancers will not exclude patients from participating in this study.
* Patients with previously documented human immunodeficiency virus (HIV) infection. HIV-positive patients are excluded from the study based on theoretical concerns regarding the effect of PS-341 on certain aspects of immune function. NF-KB is a critical T cell activation protein (including through CD40L/CD 154 stimulation) and also is involved in cytokine production. Because PS 341 effectively blocks NF-KB and therefore could reduce or block the ability of T lymphocytes and other immune cells to fight HIV, PS-341 should not be administered to HIV-positive patients. Additional experiments in animal models are being conducted to better elucidate the effects of PS-341 on HIV.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Other serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Patients who are pregnant, suspected to be pregnant, or breast-feeding.
* Patients with a known hypersensitivity to PS-341, boron, or mannitol.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Bortezomib with Carboplatin Chemotherapy | Assessed Day 21 of each 28 Day cycle, up to 4 cohorts for a total of 8 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Pedro T. Ramirez, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org